CLINICAL TRIAL: NCT05959460
Title: Validation of Maternal Recall of Exclusive Breastfeeding by the Deuterium Dilution Method: a Study in 7 Asian Countries
Brief Title: Assessing Exclusive Breastfeeding Practice
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: Pakistan Institute of Nuclear Science and Technology (PINSTECH) (Other Government); Faculty of Medicine, University of Ruhuna, Sri Lanka (Unknown); National Institute of Nutrition, Vietnam (Other Government); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); International Atomic Energy Agency (Other Government); St. John's Research Institute (Other); National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other); Research Organization for Nuclear Energy-BRIN Indonesia (Unknown); National University of Malaysia (Other); National Center for Maternal and Child Health, Mongolia (Unknown)
Responsible Party: Principal Investigator, Pattanee Winichagoon, Associate Professor Dr., Mahidol University
Other Study IDs: RAS6073
Record Dates: First submitted 2023-07-16; First posted 2023-07-25 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Exclusive Breastfeeding; Human Milk; Breast Milk
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: This is an observation study to determine exclusive breastfeeding practice. Mother-child pairs were enrolled at 3 months ± 7d and were followed-up at 6 months ± 7d. Questionnaire was administered. Then, baseline saliva samples were collected and deuterium oxide dose was administered. Then, post-dose saliva samples were collected.
  Interventions: Other: Deuterium dose-to-mother method for assessing breastfeeding

INTERVENTIONS:
Other: Deuterium dose-to-mother method for assessing breastfeeding — Exclusive breastfeeding practice was compared between maternal recall and the deuterium dose-to-mother method.

SUMMARY:
This study was a longitudinal design. The questionnaire on exclusive breastfeeding was administered and was validated against the deuterium oxide dose-to-mother technique to assess human milk intake of babies aged 3 and 6 mo.

DETAILED DESCRIPTION:
This study is a longitudinal design that aimed to assess exclusive breastfeeding (EBF) practices in Asian countries and to compare the agreement in EBF between maternal recall and the dose-to-mother technique (DTM) technique. The questionnaire on exclusive breastfeeding was administered and was validated against the deuterium oxide dose-to-mother technique to assess human milk intake of babies aged 3 and 6 mo. The study planned to recruit 30 mother-baby pairs from each participated country. The was carried out in 7 countries in Asia, namely, Indonesia, Malaysia, Mongolia, Pakistan, Sri Lanka, Thailand, and Vietnam.

Mothers were approached at child birth, to explain the project objective and obtain written informed consent. A screening questionnaire was administered to obtain the interest to participate in the study. Only mothers who intend to exclusive breastfeeding till 6 mo will be eligible for further information and sample collection. Isotope dosing of mothers and saliva sample collection were done when the baby is at 3 mo ± 1wk, when a questionnaire (validation questionnaire) was administered. A basal saliva sample was collected prior to dosing with deuterium oxide. The isotope dosing of the mother was given and saliva samples were collected (post-dose) on day 1,2,3,4 and days 13,14.

The mother-baby pairs were followed up for another sample collection at 6 mo ± 1 wk and all procedures were repeated, including a questionnaire administration, basal sample collection, deuterium oxide dose administration, and post-dose sample collection. Body weight and height/length of mothers and infants were measured. All saliva samples were analyzed by Isotope ratio mass spectrometer (IRMS) or Fourier Transform Infrared Spectroscopy (FTIR).

Quantity of breast milk intake, non milk oral intake (NMOI) and maternal body composition were determined using standard assumption and formulae developed by the International Atomic Energy Agency (IAEA). Children with NMOI ≥ 86.6 g/day were considered as non-EBF using stable isotopic DTM technique. The overall agreement of EBF classification between the recall and DTM techniques is presented using Kappa statistic with 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Mother who practice exclusive breastfeeding
* Age of mother 18 - 40 years
* Parity: no more than 3
* Baby 3 month ± 7 days
* Nutritional status Weight-for-height Z score (WHZ) > -2
* Full term baby (37 - 40 weeks)

Exclusion Criteria:

* Twin or more baby
* Low birth weight
* Baby with oedema
* Mother with fluid retention disease (kidney disease, heart disease, hypothyroidism)
* Smoking mother
* Drinking alcohol mother

Ages: 3 Months to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The participants were mother-baby pairs who were eligible according to the inclusion and exclusion criteria. There were recruited from hospitals, health clinics, or communities.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Non-milk oral intake | Jan 2016 - Dec 2020
  Quantity of non-milk oral intake (g)
Human milk intake | Jan 2016 - Dec 2020
  Quantity of milk intake (g)

SECONDARY OUTCOMES:
Body composition of mothers: total body water | Jan 2016 - Dec 2020
  Total body water in kilograms and as a percentage of body weight
Body composition of mothers: fat free mass | Jan 2016 - Dec 2020
  Fat free mass in kilograms and as a percentage of body weight
Body composition of mothers: fat mass | Jan 2016 - Dec 2020
  Fat mass in kilograms and as a percentage of body weight
Weight of infants | Jan 2016 - Dec 2020
  Body weight in kilograms
length of infants | Jan 2016 - Dec 2020
  Body length in centimeters. Weight-for-age, length-for-age, and weight-for-length z-scores were calculated based on the World Health Organization (WHO) growth standard.
Weight of mothers | Jan 2016 - Dec 2020
  Body weight in kilograms
Height of mothers | Jan 2016 - Dec 2020
  Height in centimeters. The body mass index (BMI) was calculated by dividing weight in kilograms by height in meters squared.
Body mass index of mothers | Jan 2016 - Dec 2020
  weight in kilograms divided by height in meters squared
Breastfeeding pattern | Jan 2016 - Dec 2020
  Breastfeeding pattern based on questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tippawan Pongcharoen, PhD, Study Director — Mahidol U

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tongchom W, Pongcharoen T, Judprasong K, Udomkesmalee E, Kriengsinyos W, Winichagoon P. Human Milk Intake of Thai Breastfed Infants During the First 6 Months Using the Dose-to-Mother Deuterium Dilution Method. Food Nutr Bull. 2020 Sep;41(3):343-354. doi: 10.1177/0379572120943092. Epub 2020 Aug 17. PMID 32799695
- [Background] Mulol H, Coutsoudis A. Limitations of maternal recall for measuring exclusive breastfeeding rates in South African mothers. Int Breastfeed J. 2018 May 25;13:19. doi: 10.1186/s13006-018-0159-8. eCollection 2018. PMID 29849742
- See also: https://www.iaea.org/publications/8168/stable-isotope-technique-to-assess-intake-of-human-milk-in-breastfed-infants — https://www.iaea.org/publications/8168/stable-isotope-technique-to-assess-intake-of-human-milk-in-breastfed-infants